CLINICAL TRIAL: NCT03002844
Title: EGFR-TKI With/Without Chemotherapy in NSCLC Patients With Both EGFR Mutation and BIM Deletion Polymorphism
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Director Head of Medical Oncology, Principal Investigator, Clinical Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiPH002
Record Dates: First submitted 2016-12-14; First posted 2016-12-26 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Nonsmall Cell Lung Cancer; EGFR Gene Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Drug Therapy; Pemetrexed; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EGFR-TKI and Chemotherapy (Experimental): gefitinib with pemetrexed/gemcitabine and carboplatin
  Interventions: Drug: EGFR-TKI; Drug: EGFR-TKI and Chemotherapy
- EGFR-TK Inhibitor (Experimental): Gefitinib
  Interventions: Drug: EGFR-TK Inhibitor

INTERVENTIONS:
Drug: EGFR-TK Inhibitor — EGFR-TKI (gefitinib 250mg per day)
  Other Names: gefitinib
  Arms: EGFR-TK Inhibitor
Drug: EGFR-TKI — EGFR-TKI (gefitinib 250mg per day)
  Other Names: gefitinib
  Arms: EGFR-TKI and Chemotherapy
Drug: EGFR-TKI and Chemotherapy — pemetrexed 500mg per kg q3w/gemcitabine 1000mg per kg q3w and carboplatin AUC=5 q3w
  Other Names: EGFR-TKI and pemetrexed/gemcitabine and carboplatin
  Arms: EGFR-TKI and Chemotherapy

SUMMARY:
BIM deletion polymorphism might be associated with a poor clinical response to EGFR-TKIs in patients who had NSCLC with EGFR mutations. In the study, the investigators want to use EGFR-TKI with/without chemotherapy as first line treatment in stage IIIB/IV NSCLC patients with both EGFR mutation and BIM deletion polymorphism.

DETAILED DESCRIPTION:
BIM deletion polymorphism was a poor clinical response marker to EGFR-TKIs in NSCLC patients who had EGFR mutations. In the study, the investigators want to use EGFR-TKI with chemotherapy as 1 st treatment in stage IIIB/IV NSCLC patients with both EGFR mutation and BIM deletion polymorphism.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Histologically documented, unresectable, inoperable, locally advanced, recurrent or metastatic Stage IV Non-Small Cell Lung Cancer (NSCLC)
3. Must have measurable or non-measurable disease
4. Must be able to comply with study and follow-up procedures

Exclusion Criteria:

1. Small cell, carcinoid, or mixed small cell lung cancer
2. Malignancies within 3 years except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer
3. Symptomatic or untreated brain metastases Prior systemic chemotherapy for NSCLC
4. Unstable systemic disease, including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months prior to Day 1, or serious cardiac arrhythmia requiring medication
5. History of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the patient at high risk from treatment complications
6. Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, or prior surgical procedures affecting absorption
7. Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival | up to 12 months

SECONDARY OUTCOMES:
Overall Survival | up to 24 months
Overall Response Rate | up to 12 months
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | up to 12 months
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD, PHD, Principal Investigator — Shanghai Pulmonary Hospital, Tongji University

IPD SHARING:
Plan to Share IPD: No